CLINICAL TRIAL: NCT05032664
Title: Effectiveness of Home-based Family Caregiver-delivered Aromatherapy Programme for the Management of Behavioural and Psychological Symptoms of Dementia for Older Persons With Dementia
Brief Title: Effectiveness of Home-based Aromatherapy for BPSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Siu Yin, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021.335
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Behavioural and Psychiatric Symptoms of Dementia
Keywords: BPSD; Dementia; Aromatherapy
MeSH Terms: conditions — Dementia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Home-based aromatherapy programme
  Interventions: Other: Home-based aromatherapy programme
- Control Group (Other): Wait-list control
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Home-based aromatherapy programme — 1 hour individualised face-to-face training to family caregivers, and 3 weeks aromatherapy intervention delivered by family caregivers (aromatherapy inhalation 2 times per day, each for 1 hour, using 2 drops of Lavandula angustifolia essential oil.
  Arms: Intervention Group
Other: Control Group — Wait-list control, no intervention for 3 weeks, then provide home-based aromatherapy
  Arms: Control Group

SUMMARY:
Behavioral and psychological symptoms of dementia (BPSD) is the most prominent and distressing manifestation for older persons with dementia (PWD) and caregivers. Aromatherapy was a potentially safe and effective non-pharmacological strategy in BPSD management and could provide benefits to PWD and caregivers. In Hong Kong, some Residential Care Homes for the Elderly and day care centres have provided aromatherapy service to the PWD receiving service from them. However, no such service was provided to the community-dwelling PWD living at home, which constitute a larger proportion of dementia population in HK. In addition, there is no clear implementation protocol, or formal training to the family caregivers to deliver aromatherapy to PWD in home-based setting. Therefore, this study aims to develop and evaluate the effectiveness of a home-based family caregiver-delivered aromatherapy programme for the management of BPSD.

PWD ≥ 60-year-old, with BPSD symptoms, and living at home, as well as their family caregivers will be recruited. Participants who pass the screening are randomly allocated to intervention or control group. Those in the intervention group receive home-based aromatherapy programme. Those in the control group receive no intervention for 3-week control period, and then receive home-based aromatherapy programme.

The outcome measures will be conducted at baseline and after the 3-week intervention/control period by using Chinese versions of Neuropsychiatric Inventory (CNPI), Chinese version of Dementia QoL Measure-Proxy (C-DEMQoL-Proxy), and Chinese version of Zarit Burden Interview (CZBI).

DETAILED DESCRIPTION:
Study Aim and Objectives:

This study aims to develop and evaluate the effectiveness of a home-based family caregiver-delivered aromatherapy programme for the management of BPSD.

The objectives are to evaluate the effectiveness of the programme in improving PWD's severity of BPSD symptoms and QoL, and decreasing family caregivers' distress and burden.

Study Design and Setting:

This study is a RCT with two-armed single-blinded parallel design conducted in the participants' homes.

Intervention Group: Home-based Aromatherapy Programme After baseline assessment, an evidence-based theory-driven home-based aromatherapy programme will be conducted in intervention group.

Control Group: Wait-list Control After baseline assessment, no intervention will be provided to the control group for a 3-week control period. Afterwards, individualised face-to-face training will be provided to the family caregivers, and aromatherapy materials will be provided for delivering home-based aromatherapy intervention on PWD.

Study Outcomes:

The primary outcome is the change in PWD's severity of BPSD symptoms. The secondary outcomes are the changes in PWD's QoL, and family caregivers' distress and burden.

Process Evaluation:

Process evaluation will be performed in intervention group by:

1. Skill assessment checklist is used to assess the family caregivers' competence in delivering aromatherapy.
2. Logbook is used to monitor the adherence to the programme.
3. Regular consultation with consultation record form is used to monitor the feasibility, acceptance, and any adverse effect and perceived barriers to the intervention.
4. 15-20 minutes semi-structured individual interview with an interview guide to family caregivers after intervention is used to evaluate the feasibility, acceptability, and perceived benefit and limitation of the programme.

Data Analysis Plan

Analysis of Quantitative Data:

The normality of continuous variables will be assessed by using z-test for skewness and kurtosis. Skewness and kurtosis statistics are less reliable in sample size of less than 300 because they could not adjust the standard error; therefore, z-test will be applied for normality test using skewness and kurtosis. The homogeneity of the baseline data between the intervention and control groups, and between the participants who have completed the study and those do not, will be analysed using independent-sample t-test, Mann-Whitney U test, Pearson chi-square test, or Fisher's exact test depending on the type and normality of the data. The outcome variables are expressed as continuous variables. The differential changes of outcomes between groups and across time will be evaluated by generalized estimating equation (GEE) models.

Analysis of Qualitative Data:

The qualitative data will be analysed by conventional content analysis. They will be read repeatedly to derive codes. The codes will then be sorted into different subcategories by inductive method. Then, the subcategories will be combined to form categories based on the relationships between subcategories. Finally, all the categories, subcategories and codes will be determined after discussion within the research team.

ELIGIBILITY:
Inclusion Criteria:

The PWD must satisfy the following criteria to be included in the study:

* 60 years old or above
* residing at home
* with a diagnosis of dementia of any type and stage of severity
* presenting with at least one symptom of BPSD in the previous one month before the study
* able to communicate in Cantonese or Mandarin

The caregivers must satisfy the following criteria to be included in the study:

* family members, partners, or relatives living with PWD
* provide unpaid daily care to PWD at home
* literate in Chinese and able to communicate in Cantonese or Mandarin.

Exclusion Criteria:

PWD and their family caregivers are excluded from the study if either of them have:

* allergy or discomfort after using Lavender essential oil
* other neurological or psychological diseases besides BPSD
* the following conditions: pregnancy, breastfeeding, hypotension, exacerbation of asthma, dyspnoea, epilepsy, or glucose-6-phosphate dehydrogenase deficiency
* current use of the following drugs: anticoagulant Warfarin, antiplatelet Aspirin, central nervous system depressant, or anticonvulsant
* hate the smell of Lavender or Lavender essential oil
* PWD have received aromatherapy in the past one month
* a change in family caregiver within 1 month before the study or during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change of older persons with dementia (PWD)'s severity of BPSD as assessed by CNPI | baseline, after 3-week intervention/ control period
  Chinese versions of Neuropsychiatric Inventory (CNPI) is used to assess the frequency, severity, and degree of caregiver distress of 12 domains of BPSD symptoms Each domain contains one screening question, followed by 7-9 sub-questions. If the caregivers answered 'yes' or had uncertainties in the screening question, sub-questions will be used to confirm the screening question. After confirmation, the caregivers will be asked to rate the frequency (from 1 = occasionally to 4 = very frequently) and severity (from 1 = mild to 3 = severe) of symptoms, and the degree of caregiver distress (from 0 = no distress to 5 = very severe or extreme) for that domain. The total score of each domain will be calculated by multiplying the frequency by severity. The total score for the severity of BPSD symptoms will be calculated by adding the total scores for each domain; a higher score indicates higher severity of BPSD symptoms.

SECONDARY OUTCOMES:
Change of PWD's quality of life as assessed by C-DEMQoL-Proxy | baseline, after 3-week intervention/ control period
  Chinese version of Dementia Quality of Life Measure - Proxy (DEMQoL-Proxy) is a 31-item caregiver-reported questionnaire used to measure the quality of life (QoL) of PWD by assessing the feelings, memory, and daily life. Each item is rated in a four-point Likert scale (from 1 = a lot to 4 = not at all), with a total score ranging from 31 to 124, and a higher score indicating better QoL.
Change of family caregivers' distress as assessed by CNPI | baseline, after 3-week intervention/ control period
  CNPI is used to assess the frequency, severity, and degree of caregiver distress of 12 domains of BPSD symptoms Each domain contains one screening question, followed by 7-9 sub-questions. If the caregivers answered 'yes' or had uncertainties in the screening question, sub-questions will be used to confirm the screening question. After confirmation, the caregivers will be asked to rate the frequency (from 1 = occasionally to 4 = very frequently) and severity (from 1 = mild to 3 = severe) of symptoms, and the degree of caregiver distress (from 0 = no distress to 5 = very severe or extreme) for that domain. The total score of each domain will be calculated by multiplying the frequency by severity. The total caregiver distress score will be calculated separately by adding the individual caregiver distress score for each domain; a higher score indicates higher caregiver distress
Change of family caregivers' burden as assessed by CZBI | baseline, after 3-week intervention/ control period
  Chinese version of Zarit Burden Interview (CZBI) contains 22 items to assess the subjective burden reported by the caregivers of PWD. Each item is rated by a five-point Likert scale ranging from 0 = never to 4 = nearly always for the first 21 items, and from 0 = not at all to 4 = extremely for the last item, with a total score ranging from 0 to 88, and a higher score indicating higher caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Siu Yin Li, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Individual applicants, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data contain participants' privacy

REFERENCES:
- [Derived] Li BSY, Cheung AT, Chow KM, Chan CWH. Effects of a home-based aromatherapy programme for the management of behavioural and psychological symptoms of dementia among older persons with dementia: A randomised controlled trial with process evaluation. Integr Med Res. 2025 Jun;14(2):101113. doi: 10.1016/j.imr.2024.101113. Epub 2024 Dec 2. PMID 40496446